CLINICAL TRIAL: NCT06085768
Title: A Preliminary Study on the Intervention Effect of Virtual Reality Exposure Therapy on Fear of Flying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMHC-VR-002
Record Dates: First submitted 2023-10-03; First posted 2023-10-17 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Fear of Flying; Virtual Reality Exposure Therapy
Keywords: fear of flying; virtual reality exposure therapy
MeSH Terms: conditions — Aerophobia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VRE intervention group (Experimental): The intervention group will receive 2 VR exposure interventions, once a week, and each intervention will experience 2 complete flight processes for about 90 minutes each time. A complete flight process includes: (1) waiting for the airport bus at the station, (2) check-in, security check, waiting, and boarding at the airport, (3) taxiing, taking off, cruising, landing, and leaving the aircraft during flight. Among them, the flight process requires the participant to sit on the flight seat, which takes about 24 minutes each time.
  A scale assessment and skin electrode and heart rate data collection will be conducted before and after each intervention. The participants' skin electrode and heart rate data will also be collected during the intervention. They will be followed up in the 2nd week after the intervention. Follow-up content includes scale evaluation and safety evaluation.
  Interventions: Behavioral: VRE intervention
- wait-list control group (No Intervention): The control group will receive scale assessments in weeks 1, 2, and 4, and after the waiting period, receive the same VR exposure intervention once a week for 2 weeks as the intervention group.

INTERVENTIONS:
Behavioral: VRE intervention — Virtual reality exposure therapy is a new treatment technology developed in recent years. This technology combines virtual reality technology with traditional exposure therapy, and uses virtual reality technology to present the exposure scenes required for exposure therapy. Therefore, it can break through the limitations of time and space and more intuitively display some things that are difficult to simulate in the treatment room. Scenes do not require the client to undergo treatment through imaginary exposure, thereby increasing the immersion and reality of the treatment. Over the past two decades, numerous studies have explored and proven the effectiveness of virtual exposure therapy.
  Arms: VRE intervention group

SUMMARY:
The goal of this clinical trial is to explore the efficacy of VR exposure intervention in alleviating fear of flying through a randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* The flight anxiety situations questionnaire (FAS) score is no less than 56 points (the critical value is set as two or more standard deviations higher than the average of the normal population);
* Aged between 18 and 65 years old;
* Have normal intelligence and good or corrected vision;
* No family history of any mental illness or other mental disorders other than anxiety disorder;
* Currently not receiving any treatment for phobia, including but not limited to taking psychotropic drugs (unless the dose is stable for more than 3 months, and the subject agrees to continue taking the dose throughout the study);
* Have at least 1 flight experience;

Exclusion Criteria:

* The participant cannot tolerate or adapt to VR stimulation;
* The participant was unable to immerse themselves well in the VR environment;
* Severe physical diseases and physical diseases induced by stimulation, including cardiovascular and respiratory diseases, etc.;
* Have a history of neurological diseases (such as epilepsy, cerebrovascular accident, etc.) or brain trauma or brain surgery;
* The subject suffers from a physical disease and is not in a stable treatment period (such as hyperthyroidism, visual impairment, etc.), resulting in the inability to fully participate in the experimental process;
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Flight Anxiety Situations Questionnaire(FAS) | from baseline to 4 weeks
  It was compiled by Van Gerwen et al. in 1999 to assess flight-related anxiety in different situations. It consists of 32 items rated on a 5-point scale from 1 ("Not at all anxious") to 5 ("Extremely anxious"). "), with a total score of 32-160 points. The scale consists of three subscales that assess anticipatory flight anxiety (anxiety that occurs when a person anticipates flying), in-flight anxiety, and generalized flight anxiety, with item numbers of 14, 11, and 7 respectively. This questionnaire has good reliability and validity, has established norms, can be used as a clinical measurement tool for fear of flying, is widely used in clinical practice and research, and is used as the main efficacy indicator.

SECONDARY OUTCOMES:
Flight Anxiety Modality Questionnaire(FAM) | from baseline to 4 weeks
  It was compiled by Van Gerwen et al. in 1999 and is used to measure the symptom pattern of expressing anxiety in flight situations, including a somatic pattern related to physical symptoms and a cognitive pattern related to the cognition of presence of pain, with a total of 18 items. , rated on a 5-point scale from 1 ("not at all") to 5 ("very strongly"), with a total score of 18-90. The questionnaire has good reliability and validity.
The Beck Anxiety Inventory(BAI) | from baseline to 4 weeks
  It was compiled by Aaron T. Beck et al. in 1988, there are 21 items in total. The person who fills out the form needs to select the impact of each symptom on him, using a 4-point rating, from 0 ("no impact") to 3 ("severe impact") "), the total score is the sum of all question scores, ranging from 0 to 63 points. The higher the total score, the more serious the subject's anxiety. The Chinese version of BAI has good reliability and validity and is widely used in clinical patients and the general population.
State-Trait Anxiety Inventory(STAI) | STAI-t is assessed only once at baseline. STAI-s is assessed from baseline to 4 weeks.
  It was developed by American psychologist Spielberg and others in the late 1960s. It consists of two subscales, including state anxiety subscale and trait anxiety subscale. Each subscale contains 20 items, rated on a 4-point scale from 1 ("not at all") to 4 ("very much"), with higher scores indicating higher levels of anxiety. The Chinese version of STAI has good reliability and validity, and the state anxiety consistency coefficient is 0.90.
Subjective Units of Distress(SUDs) | assessed every one minute during intervention, up to 24 hours
  It was developed by Wolpe in 1969 that measures the subjective intensity of the pain or distress an individual is currently experiencing through the individual's self-assessment of the position of the current anxiety, fear, or pain situation on the scale. It is primarily used in exposure therapy and is one of the most common scales used to assess treatment progress and how anxiety levels are reduced.
Igroup Presence Questionnaire(IPQ) | The IPQ should be assessed each time after the VRE intervention for participants with fear of flying. (at week 1, 2)
  It was compiled by Schubert et al. in 2001, with a total of 14 items and a 5-level score, including three dimensions: spatial immersion, involvement and realism. Wang Xi and others revised the Chinese version on this basis. After exploratory factor analysis, they found that the load of question 11 "How real is the virtual environment to you" was low, so it was deleted. The questionnaire has good reliability and validity.
Stimulator Sickness Questionnaire(SSQ) | The SSQ should be assessed each time after the VRE intervention for participants with fear of flying. (at week 1, 2)
  It was developed by Kennedy et al. in 1993 and is widely used in the evaluation of virtual reality systems. It is divided into three categories: eye discomfort, disorientation and nausea, including general discomfort, fatigue, headache, visual fatigue, difficulty Sixteen indicators including concentration.
Physiological indicators | from baseline to 2 weeks
  Data recording uses shimmer3 GSR biosensors, including galvanic skin response sensors, light pulse sensors (earlobes), and a notebook equipped with signal acquisition software to record the participant's galvanic skin response and heart rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China